CLINICAL TRIAL: NCT02842294
Title: Etude de Cohorte évaluant l'Impact de l'Association chimiothérapie et Bevacizumab en 1ère Ligne du Cancer Colorectal métastatique Sur la qualité de Vie Relative Des Patients. Etude COBEQOL
Brief Title: Cohort Study to Assess Impact of Chemotherapy Plus Bevacizumab on Health Related Quality of Life in First Line Metastatic Colorectal Cancer
Acronym: COBEQOL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2012/151
Record Dates: First submitted 2016-07-20; First posted 2016-07-22 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Metastatic Colorectal Cancer; Quality of Life
Keywords: bevacizumab; health related quality of life
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- irinotecan based chemotherapy: patients having a 1st line doublet chemotherapy including irinotecan
  Interventions: Drug: Bevacizumab
- oxaliplatin based chemotherapy: patients having a 1st line doublet chemotherapy including oxaliplatin
  Interventions: Drug: Bevacizumab
- triplet chemotherapy: patient having a 1st line triplet chemotherapy including oxaliplatin / irinotecan this cohort was added while primary objective was to compare doublet chemotherapy
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab

SUMMARY:
The primary aim of this french multicenter national study is to assess and compare time to quality of life score deterioration (targeted dimensions : global health, fatigue and emotional functionning of EORTC QLQC30 according to the first line chemotherapy associated with bevacizumab in metastatic colorectal patients.

ELIGIBILITY:
Inclusion Criteria:

* age> 18years
* metastatic colorectal cancer (non resectable)
* 1st chemotherapy including bevacizuman

Exclusion Criteria:

* treatment contre-indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: metastatic colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2013-05; Primary Completion 2017-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
time to health related quality of life score deterioration (targeted dimensions of EORTC QLQC30 : global health, fatigue, emotional functioning) | 1 year
  The EORTC QLQ-C30 is a questionnaire developed to assess the quality of life of cancer patients.

SECONDARY OUTCOMES:
time to health related quality of life score deterioration (non targeted dimensions of EORTC QLQC30 and CR 29) | 1 year
INT PATSAT32 | 1 year
  The EORTC IN-PATSAT32 is a 32-item satisfaction with care questionnaire to measure patients' appraisal of hospital doctors and nurses, as well as aspects of care organisation and services. It addresses technical competence, information provision, interpersonal skills, availability, waiting time, access, comfort and overall care perception
quality-adjusted life years (QALYs) using EQ5D | 1 year
Overall survival | 2 years
Progression Free Survival | 1 year
treatment preference | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Franck Bonnetain, PhD, Study Director — University Hospital of Besancon
Locations (1):
- CHRU Besançon, Besançon, Franche Comté, France

REFERENCES:
- See also: Related Info — http://www.umqvc.org/en/index.html